CLINICAL TRIAL: NCT05102318
Title: Clinical and Radiographic Evaluation of Mineral Trioxide Aggregate and Biodentine as Pulp Medicaments in Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: British University In Egypt (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Magdy, Director, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ain Shams University
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Pulp Disease, Dental
Keywords: Direct pulp capping, Partial Pulpotomy, and Pulpotomy
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Direct Pulp Capping with Biodentine (Experimental): Direct Pulp Capping with Biodentine
  Interventions: Procedure: Direct Pulp Capping
- Partial Pulpotomy with Biodentine (Experimental): Partial Pulpotomy with Biodentine
  Interventions: Procedure: Partial Pulpotomy
- Pulpotomy with Biodentine (Experimental): Pulpotomy with Biodentine
  Interventions: Procedure: Pulpotomy
- Direct Pulp Capping with MTA (Experimental): Direct Pulp Capping with MTA
  Interventions: Procedure: Direct Pulp Capping
- Partial Pulpotomy with MTA (Experimental): Partial Pulpotomy with MTA
  Interventions: Procedure: Partial Pulpotomy
- Pulpotomy with MTA (Experimental): Pulpotomy with MTA
  Interventions: Procedure: Pulpotomy

INTERVENTIONS:
Procedure: Direct Pulp Capping — Direct Pulp Capping
  Arms: Direct Pulp Capping with Biodentine; Direct Pulp Capping with MTA
Procedure: Partial Pulpotomy — Partial Pulpotomy
  Arms: Partial Pulpotomy with Biodentine; Partial Pulpotomy with MTA
Procedure: Pulpotomy — Pulpotomy
  Arms: Pulpotomy with Biodentine; Pulpotomy with MTA

SUMMARY:
The aim of the present study is to evaluate Mineral Trioxide Aggregate and Biodentine in direct pulp capping, partial pulpotomy, and pulpotomy in primary molars.

DETAILED DESCRIPTION:
Screening of patients will continue until the target population is achieved. Identifying and recruiting potential subjects is achieved through patient database in Pediatric Dentistry department.

A total of 150 primary molars from healthy subjects will be selected from the Pediatric Dentistry and Dental Public Health outpatient clinic, Faculty of Dentistry, Ain shams University.

Subjects will be assigned randomly into two different treatment groups as follows:

MTA Group (1):

1. Group 1(A): MTA Direct Pulp Capping. (n=25)
2. Group 1 (B): MTA Partial Pulpotomy. (n=25)
3. Group 1 (C): MTA Complete Pulpotomy. (n=25)

BiodentineTM Group (2):

1. Group 2(A): BiodentineTM Direct Pulp Capping. (n=25)
2. Group 2 (B): BiodentineTM Partial Pulpotomy. (n=25)
3. Group 2 (C): BiodentineTM Complete Pulpotomy. (n=25)

ELIGIBILITY:
Inclusion Criteria:

* No clinical symptoms or history implying irreversible pulpitis such as spontaneous pain, or pain persisting after stimuli removal.
* Absence of periapical or interadicular radiolucencies, inflammatory root resorption, sinus tract or gingival abscess.

Exclusion Criteria:

* Children who are extremely uncooperative and difficult to manage.
* Children suffering from any physically or mentally disability that will complicate the treatment: Special Health Care needs (SHCN).
* Teeth of poor prognosis due to presence of an abscess or a sinus, mobility, advanced bone or root resorption or Non-Restorable teeth.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Is to evaluate the clinical and radiographic success rates of Mineral Trioxide Aggregate and Biodentine in direct pulp capping, partial pulpotomy, and pulpotomy in primary molars. | 18 months
  Is to evaluate the clinical and radiographic success rates of Mineral Trioxide Aggregate and Biodentine in direct pulp capping, partial pulpotomy, and pulpotomy in primary molars.

CONTACTS AND LOCATIONS:
Overall Officials: Noha Kabil, Professor, Study Director — British University In Egypt
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No